CLINICAL TRIAL: NCT06697015
Title: Comparative Effects of Pendulum Exercise and Serratus Punch Exercises on Rotator Cuff Pain and Disability in Badminton Players
Brief Title: Comparative Effects of Pendulum Exercise and Serratus Punch Exercises on Rotator Cuff Pain in Badminton Players
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0430
Record Dates: First submitted 2024-11-18; First posted 2024-11-20 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Sports Physical Therapy
Keywords: Rotator Cuff Injuries; Shoulder Pain; Badminton Injuries; Rehablitation
MeSH Terms: conditions — Rotator Cuff Injuries; Shoulder Pain

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant
Masking Description: The participants are blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pendulum Exercises (Active Comparator): Eighteen participants will perform pendulum exercises, which involve gently swinging the arm to relax shoulder muscles and improve mobility. This low-impact exercise is intended to alleviate tension and increase circulation in the rotator cuff, making it ideal for early-stage shoulder rehabilitation.
  Interventions: Other: Pendulum Exercises
- Serratus Punch Exercises (Active Comparator): Eighteen participants will engage in serratus punch exercises, extending the arm in a controlled punching motion to strengthen the serratus anterior muscle. This exercise promotes shoulder stability and supports rotator cuff function, aiming to reduce pain and improve shoulder control.
  Interventions: Other: Serratus Punch Exercises

INTERVENTIONS:
Other: Pendulum Exercises — In this group, 18 participants will perform pendulum exercises, which involve leaning forward and allowing the affected arm to hang down, swinging it gently in small circular or side-to-side motions. This exercise is designed to enhance shoulder mobility and promote relaxation of the rotator cuff muscles without straining the shoulder joint. The pendulum movement helps improve circulation and relieve tension in the shoulder area, making it a suitable intervention for individuals experiencing rotator cuff pain.
  Arms: Pendulum Exercises
Other: Serratus Punch Exercises — In this group, 18 participants will engage in serratus punch exercises, focusing on strengthening the serratus anterior muscle. Participants will perform a punching motion by extending the arm forward while maintaining shoulder stability. This exercise activates the shoulder muscles to enhance scapular control, supporting the rotator cuff and improving overall shoulder function. The goal is to build strength in the stabilizing muscles, which can help alleviate pain and enhance mobility in participants suffering from rotator cuff issues.
  Arms: Serratus Punch Exercises

SUMMARY:
This study will compare the effects of two exercise interventions, pendulum exercises and serratus punches, on rotator cuff pain and injury in badminton players. Using a randomized clinical trial with participants from local clubs, the research will evaluate pain levels, range of motion, and shoulder function after a set period of regular, supervised exercises. The results aim to provide evidence-based insights for effective rehabilitation programs tailored to badminton athletes, supporting better recovery and injury prevention.

DETAILED DESCRIPTION:
Rotator cuff pain and disability is typical among badminton players because of the dull movements associated with the game. These wounds can prompt critical torment and practical limits, influencing the players' exhibition and prosperity. The focal point of this exploration project is to think about the impacts of two different activity mediations, pendulum activities and serratus punch works, on rotator sleeve agony and injury in badminton players. Understanding the similar adequacy of these activities will contribute essential knowledge to improving designated restoration programs for badminton competitors, further developing their recuperation results and forestalling future wounds.

This exploration will utilize a randomized clinical preliminary plan to research the similar impacts of pendulum activities and serratus punch practices on rotator sleeve agony and injury in badminton players. Members will be selected from neighborhood badminton clubs, and consideration measures will include people with an analyzed or self-revealed history of rotator sleeve torment. The chosen members will be arbitrarily allotted to the pendulum or the serratus punch practice bunch. The mediation time frame will traverse a predefined span, during which members will routinely participate in their doled-out practice. Result estimates will incorporate torment levels, scope of movement, and practical appraisals of the rotator sleeve. Factual examinations will be directed to consider the viability of the two activity mediations and their effect on rotator sleeve agony and injury in badminton players. The consequences of this study are to illuminate proof-based restoration systems customized explicitly for the badminton populace, adding to the enhancement of player well-being and execution.

ELIGIBILITY:
Inclusion Criteria:

* Badminton players aged 15 to 30 years.
* Individuals with self-reported rotator cuff pain or discomfort
* Clinically diagnosed rotator cuff pain or discomfort.
* Individuals with Rotator Cuff Injury.

Exclusion Criteria:

* Previous shoulder surgeries or fractures.
* Chronic shoulder conditions unrelated to rotator cuff issues.
* Inability to perform the prescribed exercises due to other musculoskeletal or medical conditions.
* Patients with shoulder dislocation.
* Patients with swelling on shoulder.

Ages: 15 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 36 (Actual)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-01-20 (Estimated); Study Completion 2025-01-30 (Estimated)

PRIMARY OUTCOMES:
DASH Score | 10 MONTHS
  The Disabilities of the Arm, Shoulder and Hand (DASH) score is a self-reported questionnaire that measures the disability and symptoms related to upper extremity conditions. It consists of 30 items assessing difficulties in daily activities and the presence of pain. Scores range from 0 to 100, where 0 indicates no disability and 100 indicates maximum disability. The DASH score is useful for evaluating functional status, tracking treatment outcomes, and guiding rehabilitation in patients with arm, shoulder, and hand issues.
Oxford Shoulder Score | 10 months
  The Oxford Shoulder Score (OSS) is a patient-reported outcome measure that assesses shoulder pain and disability. It includes 12 items focusing on pain levels and functional limitations related to daily activities. Scores range from 0 to 48, with higher scores indicating better shoulder function. The OSS is commonly used in clinical practice and research to evaluate treatment outcomes for shoulder conditions, providing valuable insights into the patient's perspective on their shoulder health
Range of motion | 10 months
  The shoulder's range of motion will be measured using a goniometer to assess specific movements such as flexion, extension, abduction, and internal/external rotation. Assessments will be conducted at baseline and after the intervention to evaluate improvements in mobility, providing objective data on the effectiveness of the exercise interventions for participants with rotator cuff pain.

CONTACTS AND LOCATIONS:
Overall Officials: Wafa Abid, DPT, Principal Investigator — Riphah International University
Locations (1):
- Pakistan Sports Board, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aicale R, Tarantino D, Maffulli N. Overuse injuries in sport: a comprehensive overview. J Orthop Surg Res. 2018 Dec 5;13(1):309. doi: 10.1186/s13018-018-1017-5. PMID 30518382
- [Background] Atroshi I, Gummesson C, Andersson B, Dahlgren E, Johansson A. The disabilities of the arm, shoulder and hand (DASH) outcome questionnaire: reliability and validity of the Swedish version evaluated in 176 patients. Acta Orthop Scand. 2000 Dec;71(6):613-8. doi: 10.1080/000164700317362262. PMID 11145390
- [Background] Nikolaidou O, Migkou S, Karampalis C. Rehabilitation after Rotator Cuff Repair. Open Orthop J. 2017 Feb 28;11:154-162. doi: 10.2174/1874325001711010154. eCollection 2017. PMID 28400883
- [Background] Couppe C, Thorborg K, Hansen M, Fahlstrom M, Bjordal JM, Nielsen D, Baun M, Storgaard M, Magnusson SP. Shoulder rotational profiles in young healthy elite female and male badminton players. Scand J Med Sci Sports. 2014 Feb;24(1):122-8. doi: 10.1111/j.1600-0838.2012.01480.x. Epub 2012 May 22. PMID 22616686
- [Background] Pardiwala DN, Subbiah K, Rao N, Modi R. Badminton Injuries in Elite Athletes: A Review of Epidemiology and Biomechanics. Indian J Orthop. 2020 Mar 10;54(3):237-245. doi: 10.1007/s43465-020-00054-1. eCollection 2020 May. PMID 32399141
- [Background] Cejudo A. Risk Factors for, and Prediction of, Shoulder Pain in Young Badminton Players: A Prospective Cohort Study. Int J Environ Res Public Health. 2022 Oct 12;19(20):13095. doi: 10.3390/ijerph192013095. PMID 36293672
- [Background] Padua R, Padua L, Ceccarelli E, Romanini E, Zanoli G, Amadio PC, Campi A. Italian version of the Disability of the Arm, Shoulder and Hand (DASH) questionnaire. Cross-cultural adaptation and validation. J Hand Surg Br. 2003 Apr;28(2):179-86. doi: 10.1016/s0266-7681(02)00303-0. PMID 12631494
- [Background] Hickey D, Solvig V, Cavalheri V, Harrold M, Mckenna L. Scapular dyskinesis increases the risk of future shoulder pain by 43% in asymptomatic athletes: a systematic review and meta-analysis. Br J Sports Med. 2018 Jan;52(2):102-110. doi: 10.1136/bjsports-2017-097559. Epub 2017 Jul 22. PMID 28735288